CLINICAL TRIAL: NCT05281692
Title: Prospective, Non-Randomized, Parallel Assignment and Single Site Comparison of EPM-IX to Currently Used Specimen Transportation and Extraction Devices
Brief Title: Comparison of EPM-IX to Currently Used Specimen Transportation and Extraction Devices ( CGI-EPM-IX )
Acronym: CGI-EPM-IX
Status: Completed | Type: Observational
Sponsor: Convergent Genomics, Inc. (Network)
Responsible Party: Sponsor
Other Study IDs: CGI-EPM-IX
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: SARS-CoV-2
Keywords: EPM-IX; Covid-19; SARS-CoV-2; Nasopharyngeal swab; Med Schenker's STM viral media
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EPM-IX is a clinical specimen collection medium that inactivates pathogens, preserves nucleic acids, and integrates DNA/RNA purification. EPM-IX eliminates the need for additional extraction reagents or kits and purifies DNA/RNA from the entire sample to enable optimal test performance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive: Enhanced Preservation Media (EPM-IX)
  Interventions: Diagnostic Test: Enhanced Preservation Media (EPM-IX)
- Control: Med Schenker's STM viral media
  Interventions: Diagnostic Test: Enhanced Preservation Media (EPM-IX)

INTERVENTIONS:
Diagnostic Test: Enhanced Preservation Media (EPM-IX) — EPM-IX is a clinical specimen collection medium that inactivates pathogens, preserves nucleic acids, and integrates DNA/RNA purification. EPM-IX eliminates the need for additional extraction reagents or kits and purifies DNA/ RNA from the entire sample to enable optimal test performance.

SUMMARY:
This is a research study to evaluate the clinical utility of the Enhanced Preservation Media with Integrated Extraction (EPM-IX)

DETAILED DESCRIPTION:
This is a minimal risk study where patients at UroPartners Urology Group will consent to SARS-CoV-2 nasopharyngeal swab testing using both, a standard of care test with standard Viral Transport Medium and a second test using Convergent Genomics' proprietary Enhanced Preservation Media (EPM-IX). Subjects will self-swab each nostril during their medical appointment at UroPartners. UroPartners designated staff with then send the collection kits out for testing. Clinical information will be collected that includes age, gender, race, ethnicity and history of cancer. All of these data points will be anonymized.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥18 years of age
* Subject is a current patient at UroPartners and is willing to be tested for Covid- 19 during a routine visit
* Subject must be able to understand and willingly provide informed consent

Exclusion Criteria:

* Cannot provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female subjects ≥ 18 years of age who are being tested for COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Comparison of Diagnostic Performance | At the time of inclusion
  Comparison of diagnostic performances (sensitivity, specificity, and predictive values) of EPM-IX vs Med Schenker's STM viral media with detection of SARS-CoV-2 infection.

SECONDARY OUTCOMES:
Comparison of Lab Processing | At the time of inclusion
  Comparison of Lab processing time with accessioning and processing of an EPM-IX tube compared to with Med Schenker's STM viral media
Quantitative PCR CT-values | At the time of inclusion
  Quantitative PCR CT-values (of internal control and target gene levels) using EPM-IX vs Med Schenker's STM viral media
Difference in case rate or detection of viral load samples observed | At the time of inclusion
  Difference in case rate or detection of viral load samples observed between EPM-IX and Med Schenker's STM viral media

CONTACTS AND LOCATIONS:
Overall Officials: Paul Yonover, MD, Principal Investigator — UroPartners, LLC
Locations (1):
- UroPartners Urology Group, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided